CLINICAL TRIAL: NCT02543775
Title: Sentinel Lymph Node Detection in Early Cervical Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 09-1003-CE
Record Dates: First submitted 2015-06-02; First posted 2015-09-07 (Estimated); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Cervical Cancer
Keywords: Cervical Cancer; Sentinel Lymph Node; Lymphadenectomy
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sentinel lymph node mapping (Experimental): Patients who consent to the study will have preoperative and intraoperative SLN mapping performed. This will include injection of a radioisotope (Technetium 99) into the cervix and imaging (SPECT/CT) at Nuclear Medicine in the morning prior to surgery in an effort to identify the lymph node basin containing the sentinel nodes. Intraoperatively, blue dye will also be injected into the cervix to aid in location of the sentinel nodes.
  Interventions: Procedure: Preoperative and intraoperative SLN Mapping

INTERVENTIONS:
Procedure: Preoperative and intraoperative SLN Mapping — Patients will undergo preoperative SLN mapping, which includes an injection of a radiocolloid and lymphosinctogram and SPECT/CT. Patients will also receive an intraoperative injection of blue dye. A handheld probe will be utilized to detect radiolabelled or "hot" nodes and direct visualization will identify blue nodes which will be labelled "Sentinel Nodes" and sent to pathology for intraoperative frozen section.

SUMMARY:
The primary objective of this study is to determine the feasibility of detecting the sentinel lymph node (SLN) in patients with early invasive cervical cancer using a combined radioisotope and blue dye technique.

The investigators hypothesize that the sentinel lymph node (first node draining the tumour/cervix) for early stage cervical cancer represents the status of the regional lymph node basin (pelvic lymph nodes) and identification of a negative SLN would negate the need for complete pelvic lymphadenectomy.

DETAILED DESCRIPTION:
Cancers of the cervix that are small and appear to be contained in the cervix (early stage) have up to 20 percent chance of having pelvic lymph nodes involved. The standard therapy is removal of the uterus and cervix (radical hysterectomy) and removal of all pelvic lymph nodes for all women with early stage cervical cancer. This procedure can be associated with significant intraoperative and postoperative complications including increased risk of damage to blood vessels and nerves in the pelvic region (leading to bladder, bowel and sexual dysfunction) as well as lymphedema (swelling, particularly in the legs) associated with significant pelvic lymph tissue removal.

The objective of this study is to find a way to accurately identify the first lymph node that drains the tumour/cervix (SLN). If this SLN is correctly identified, and it's status (positive or negative for malignancy) is representative of the entire lymph node basin, a complete node dissection could be avoided. This could benefit many women with early stage cervical cancer, as a minority actually have evidence of disease in the nodes after surgery (between 5-20%) and limited lymph node sampling could prevent the associated complications of a full pelvic lymph node dissection.

This is a prospective cohort study. The population to be studied is patients with newly diagnosed early stage cervical cancer undergoing primary surgical intervention including radical hysterectomy and bilateral pelvic lymphadenectomy. On the morning of surgery, preoperative injection of a radiolabeled colloid will be performed in the Nuclear Medicine Department followed by SPECT/CT to visualize the radiolabelled dye. Patients will then be taken to the operating room for their planned procedure. After initiation of general anesthesia, blue dye will be injected into the patient's cervix. The surgery will proceed and all lymph nodes that are "blue" and/or "hot" will be removed surgically, their anatomic location and laterality documented and sent for frozen section intraoperatively. The radical hysterectomy or radical trachelectomy and complete systematic bilateral pelvic lymphadenectomy will then be performed. The SLN status reported by the pathologist based on the frozen section will be compared to the status of the other nodes removed after complete lymphadenectomy and reported in the final pathology report (after formalin fixation and paraffin embedding). All data on these patients will be prospectively collected.

This protocol will determine the feasibility of SLN mapping in women with early stage cervical cancer. The primary outcomes will be to measure the rate of detection of SLN using the combination of radiolabelled and blue dye (unilateral and bilateral detection rates will be reported) as well as the sensitivity and specificity of this technique, based on assessing how well the intraoperative reading of SLN frozen section corresponds with the final pathology lymph node status after examining all lymph nodes removed by complete pelvic lymphadenectomy.

In addition, the investigators will assess the usefulness of preoperative SPECT/CT in identifying SLN and whether this modality accurately identifies the lymph node basin containing SLN compared to conventional lymphoscintigram.

ELIGIBILITY:
Inclusion Criteria:

1. Women with invasive adenocarcinoma or squamous cell carcinoma of the cervix
2. Stages 1A1 (+LVSI), 1A2 and 1B1 (< 4 cm)
3. If CT, MRI or PET have been performed preoperatively there must be no clear evidence of metastatic disease and/or parametrial involvement.
4. Patients who have signed an approved informed consent.
5. Patients who will undergo surgery that includes a radical hysterectomy and/or radical trachelectomy and bilateral lymphadenectomy via laparotomy, laparoscopy or robotic-assisted.

Exclusion Criteria:

1. Patients with known allergy to triphenylmethane compounds
2. Pregnant patient
3. Patients with previous retroperitoneal surgery
4. Patients with previous history of pelvic/abdominal radiation
5. Patients with recurrent cervical cancer
6. Any patient treated with neoadjuvant chemotherapy and/or radiation

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Sensitivity of sentinel lymph node (SLN) detection in patients with early invasive cervical cancer using a combined radioisotope and blue dye technique. | Three years

SECONDARY OUTCOMES:
SLN status correspondence with the overall pelvic lymph node positivity (specificity) as determined by lymphadenectomy (gold standard). | Three years

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Ferguson, MD, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada